CLINICAL TRIAL: NCT05551195
Title: A Multicenter, Randomized, Double-Blind, Controlled Study Evaluating the Efficacy and Safety of a Digital Therapeutic as an Adjunct to Treatment as Usual Among Women With Mild to Moderate Postpartum Depression
Brief Title: [Study Evaluating the Efficacy and Safety of a Digital Therapeutic as an Adjunct to TAU in Postpartum Depression]
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Internal company decision
Sponsor: Woebot Health (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WB001-001
Record Dates: First submitted 2022-09-19; First posted 2022-09-22 (Actual); Results first posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-01

CONDITIONS: Postpartum Depression
Keywords: Postpartum Depression; PPD; Postpartum Depression Treatment; PPD Treatment; Smartphone application; Digital therapeutic
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Intervention Model Description: 1:1 randomization
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- WB001 with adjunctive Treatment as Usual (Other): Participants randomized to the WB001 + TAU group will be asked to download and use the study application.
  Interventions: Device: WB001
- Educational Control (ED001) with adjunctive Treatment as Usual (Other): Participants randomized to the ED001 + TAU group will be asked to download and use the study application.
  Interventions: Device: ED001

INTERVENTIONS:
Device: WB001 — WB001 is a digital therapeutic for postpartum depression.
  Arms: WB001 with adjunctive Treatment as Usual
Device: ED001 — ED001 is a digital therapeutic for postpartum depression.
  Arms: Educational Control (ED001) with adjunctive Treatment as Usual

SUMMARY:
This study evaluates the efficacy of two digital therapeutics, WB001 and ED001, on depressive symptoms among women diagnosed with postpartum depression.

DETAILED DESCRIPTION:
This randomized, double-blind, controlled trial evaluates the efficacy and safety of 8 weeks of treatment of two digital therapeutics in a population of women with mild to moderate postpartum depression. Patients will be referred by an obstetrician, pediatrician, or other healthcare professional, or by other digital and site based recruitment methods and, if interested, will complete the pre-screening process. Those confirmed as eligible will be scheduled to attend a screening/baseline onsite visit. Eligible participants will be randomized to one of the two groups and will receive instructions on downloading and using the smartphone application to which they were randomized. Participants will use the app as instructed and will attend telehealth visits to complete assessments for the primary and safety endpoints at Weeks 4 and 8 (EOT).

ELIGIBILITY:
Inclusion Criteria:

1. Must have primary residence in the United States
2. Must be ≤ 92 days postpartum
3. Must be women aged 22-45 years who had onset of a major depressive episode any time during pregnancy or within 4 weeks following delivery
4. Must own or have regular access to a smartphone (Android or iOS smartphone with a recent, supported operating system), and has reliable Wi-Fi access or sufficient data plan to engage with assigned treatment condition for the duration of the study
5. Participants must have current mild-moderate depression as measured by the HAMD-6 score >7 and <13 at screening
6. Participant must have a form of TAU, defined as clinician supervised outpatient care management and includes follow-up visits, medication, psychotherapy, or some combination thereof
7. TAU must be regularly scheduled or stable for at least 4 weeks prior to baseline (BL) visit

Exclusion Criteria:

1. Gestation less than 28 weeks
2. HAMD-6 score ≤7 or ≥13 (severe depression) at screening
3. Currently pregnant or plans to become pregnant within the next 8 weeks
4. History of drug and/or alcohol use disorder within the past 12 months
5. Lifetime history of suicide attempt or ideation with a plan and intent to harm oneself during the current episode of PPD
6. Current or lifetime psychosis
7. Current or lifetime history of schizophrenia, schizoaffective disorder, bipolar disorder, and/or homicidal or infanticidal ideation
8. History of antidepressant treatment with ketamine/esketamine, electroconvulsive therapy, vagal nerve stimulation, or a deep brain stimulation device
9. History of treatment-resistant depression (TRD)
10. Fetal demise within the past 18 months

Ages: 22 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2022-11-16 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-05-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Woebot Investigational Site, Lafayette, California
  - Woebot Investigational Site, Santa Ana, California
  - Woebot Investigational Site, DeLand, Florida
  - Woebot Investigational Site, Miami Lakes, Florida
  - Woebot Investigational Site, Seminole, Florida
  - Woebot Investigational Site, Decatur, Georgia
  - Woebot Investigational Site, Glen Oaks, New York
  - Woebot Investigational Site, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | WB001 With Adjunctive Treatment as Usual | Educational Control (ED001) With Adjunctive Treatment as Usual
Started | 1 | 6
Completed | 1 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | WB001 With Adjunctive Treatment as Usual | Educational Control (ED001) With Adjunctive Treatment as Usual | Total
Number analyzed (Participants) | 1 | 6 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 6 | 7
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 6 | 7
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 1 | 4 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 1 | 4 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States: New York (Northeast) | 1 | 4 | 5
  United States: Florida (Southeast) | 0 | 1 | 1
  United States: California (West) | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Rating Scale for Depression (HAM-D)
Description: Measure of depression. This is a 6-item questionnaire, where total scores range from 0 to 22, with higher scores indicating greater severity of depression.
Time Frame: Change from Baseline to Post-treatment at Week 8
Population: One participant missing data at Week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WB001 With Adjunctive Treatment as Usual | Educational Control (ED001) With Adjunctive Treatment as Usual
Number analyzed (Participants) | 1 | 5
score on a scale | 0 (0) | -5.4 (3.36)

2. Secondary Outcome: Edinburgh Postpartum Depression Scale (EPDS)
Description: Measure of postpartum depression. A 10-item self-report questionnaire that assesses depression criteria and yields a total score from 0 to 30 where higher scores denote greater depression.
Time Frame: Change Baseline to Post-treatment at Week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WB001 With Adjunctive Treatment as Usual | Educational Control (ED001) With Adjunctive Treatment as Usual
Number analyzed (Participants) | 1 | 6
score on a scale | 0 (0) | -6.83 (6.37)

3. Secondary Outcome: Patient Health Questionnaire (PHQ-9)
Description: Measure of depression. A 9-item self-report questionnaire where total scores range from 0 to 27, with higher scores indicating greater levels of depression
Time Frame: Change Baseline to Post-treatment at Week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WB001 With Adjunctive Treatment as Usual | Educational Control (ED001) With Adjunctive Treatment as Usual
Number analyzed (Participants) | 1 | 6
score on a scale | -3 (0) | -8.17 (6.18)

4. Secondary Outcome: Generalized Anxiety Disorder Questionnaire (GAD-7)
Description: Measure of anxiety. A 7-item brief self-report questionnaire, where total score range is between 0-21, with higher scores indicate greater levels of anxiety.
Time Frame: Change from Baseline to Post-treatment at Week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WB001 With Adjunctive Treatment as Usual | Educational Control (ED001) With Adjunctive Treatment as Usual
Number analyzed (Participants) | 1 | 6
score on a scale | 1 (0) | -6.33 (2.88)

5. Secondary Outcome: Mother-to-Infant Bonding Scale (MIBS)
Description: Measure of mother-infant bond. An 8-item self-report questionnaire, where total scores range from 0 to 24, with lower scores indicating good bonding.
Time Frame: Change from Baseline to Post-treatment at Week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WB001 With Adjunctive Treatment as Usual | Educational Control (ED001) With Adjunctive Treatment as Usual
Number analyzed (Participants) | 1 | 6
score on a scale | -2 (0) | 0.17 (2.40)

6. Secondary Outcome: Clinical Global Impressions Scale - Severity of Illness (CGI-S)
Description: Measure of overall severity of current clinical presentation and symptomatology. A single item, 7-point Likert scale on which the investigator will rate patients' severity of illness based on clinical interviews and assessments relative to their experience with other patients with the same diagnosis. Responses include 0 (not assessed) and range from 1 (Normal, not at all ill) to 7 (Among the most extremely ill).
Time Frame: Change Baseline to Post-treatment at Week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WB001 With Adjunctive Treatment as Usual | Educational Control (ED001) With Adjunctive Treatment as Usual
Number analyzed (Participants) | 1 | 6
score on a scale | 0 (0) | -1.50 (0.84)

7. Secondary Outcome: Clinical Global Impressions Scale - Global Improvement (CGI-I)
Description: Measure of improvement. A single item, 7-point Likert scale that assesses the overall improvement in patients' condition at the end of treatment. The investigator will rate whether the participant's total improvement was due entirely to the intervention. Responses include 0 (not assessed) and range from 1 (very much improved) to 7 (very much worse).
Time Frame: Change from Mid-treatment at Week 4 to Post-treatment at Week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WB001 With Adjunctive Treatment as Usual | Educational Control (ED001) With Adjunctive Treatment as Usual
Number analyzed (Participants) | 1 | 6
score on a scale | 0 (0) | -1.17 (0.98)

8. Secondary Outcome: Patient Global Impression Scale (PGI)
Description: Measure of change in clinical status. A single item scale based on the CGI and adapted to the patient that mainly measures change in clinical status (PGI-C) but can also measure disease severity (PGI-S) or disease improvement (PGI-I). PGI-S responses for current illness severity range from "I Feel Fine (1)" to "I Feel Extremely Ill (4)". PGI-C responses range from "Very Much Improved (1) to "Very Much Worse (7)" since starting the trial. For both scales, lower scores indicate better outcomes.
Time Frame: PGI-S: Change from Baseline to Post-treatment at Week 8; PGI-C: Change from Mid-treatment at Week 4 to Post-treatment at Week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WB001 With Adjunctive Treatment as Usual | Educational Control (ED001) With Adjunctive Treatment as Usual
Number analyzed (Participants) | 1 | 6
score on a scale
  PGI-S | 1 (0) | -0.67 (1.21)
  PGI-C | 1 (0) | -1 (0.63)

9. Secondary Outcome: Client Satisfaction Questionnaire (CSQ-8)
Description: An 8-item measure used to assess client's satisfaction with treatment.Total scores range from 8-32, with high scores indicating greater satisfaction with the treatment.
Time Frame: Post-treatment at Week 8
Population: One participant did not complete the CSQ-8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WB001 With Adjunctive Treatment as Usual | Educational Control (ED001) With Adjunctive Treatment as Usual
Number analyzed (Participants) | 1 | 5
score on a scale | 17 (0) | 29 (4.64)

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: Systematic assessment of adverse events included Principal Investigator assessment as well as unsolicited participant reports.
Arm/Group | WB001 With Adjunctive Treatment as Usual | Educational Control (ED001) With Adjunctive Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/6
Other Adverse Events (participants affected / at risk) | 0/1 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-03): https://cdn.clinicaltrials.gov/large-docs/95/NCT05551195/Prot_SAP_000.pdf